CLINICAL TRIAL: NCT04808921
Title: Rapid Diagnostic Test for Detection of SARS-CoV-2 Antigen
Brief Title: Performance Evaluation of SARS-COV-2 (Covid-19) Antigen Rapid Test
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: As of 11 Oct 2021, IRB oversight for site is terminated. We no longer have IRB Approval to conduct this study.
Sponsor: Sky Medical Supplies & Equipments, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SKYCOV001
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV-2; Covid-19; Coronavirus
Keywords: POC; Antigen
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to validate the performance of the SARS-CoV-2 Antigen Test bioassay for rapid detection of infection when using a nasopharyngeal swab. A prospective randomized and blinded study to evaluate a rapid point of care bioassay for the detection of virus particles compared with the currently validated RT-PCR detection standard. Nasopharyngeal samples will be collected along with the current standard of care collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- SARS-CoV-2 Antigen Rapid Test (Experimental): The same group of patients participated in two arms of the study, one arm was for obtaining data on the rapid antigen test for COVID-19, the comparator arm was to obtain data from the RT-PCR
  Interventions: Diagnostic Test: Xiamen Wiz Biotech Co., Ltd. SARS-CoV-2 Antigen Rapid Test

INTERVENTIONS:
Diagnostic Test: Xiamen Wiz Biotech Co., Ltd. SARS-CoV-2 Antigen Rapid Test — Rapid Antigen diagnostic device performance comparative to RT-PCR

SUMMARY:
The SARS-CoV-2 Antigen Rapid Test is a bioassay intended for rapid point-of-care detection of the SARS-CoV-2 virus. Performance of the SARS-CoV-2 Antigen Rapid Test assay will be assessed by comparison to a reference method.

DETAILED DESCRIPTION:
The clinical performance of the SARS-CoV-2 Antigen Rapid test was evaluated in a prospective clinical study conducted at a single (1) CLIA waiver investigational site in Miami, Florida, U.S. Consenting patients of any age, gender, or race/ethnicity who presented at the test site with COVID-19 like symptoms during the 2021 COVID-19 season were sequentially enrolled and tested. Five (5) minimally trained operators with little laboratory experience and who received no training on use of the SARS-CoV-2 Antigen Rapid test and were, therefore, representative of the intended users performed the study test evaluations.

A subject's participation in this study will consist of a single visit. Following the completion of the informed consent process and a review of Inclusion/Exclusion criteria to determine eligibility, each subject will receive a unique study identification number.

ELIGIBILITY:
Inclusion Criteria:

1. Up to 200 subjects will be screened, consented, and enrolled to obtain a minimum of 60 eligible candidates. In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of informed consent
2. Subject is a suspected case of COVID-19 by clinical criteria: a patient with acute respiratory tract infection (sudden onset of at least one of the following: cough, fever, shortness of breath, fatigue, decreased appetite, myalgia) AND with no other etiology that fully explains the clinical presentation, with or without a history of close contact with a confirmed or probable COVID-19 case in the 14 days prior to onset of symptoms.
3. Subject is an appropriate candidate for Nasopharyngeal sample collection. d/. Subject is willing to provide nasopharyngeal swab samples.

Exclusion Criteria:An individual who meets the following criterion will be excluded from participation in this study:

1. Individuals who present with 10 or greater days of COVID-19 Related Symptoms, (Fever, Cough, Fatigue, Decreased Appetite, Shortness of Breath, Myalgia) or post-defervescence and/or convalescence.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Percent Positive Agreement and Negative Percent Agreement | 30 days
  Calculate the performance of the antigen test compared to PCR using nasopharyngeal swab samples

CONTACTS AND LOCATIONS:
Overall Officials: Jorge P Amaya, M.D, Principal Investigator — D&H National Research Centers INC
Locations (1):
- D&H National Research Centers INC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No